CLINICAL TRIAL: NCT05792839
Title: Concomitant Abdominoplasty with Ventral Hernia Repair Versus Ventral Hernioplasty . a Randomized Comparative Prospective Study.
Brief Title: Abdominoplasty with Ventral Hernia Repair Versus Hernioplasty .
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mark Natey Abdo Barsom, Resident at general and laparoscopic surgery department , assiut university hospital., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Abdominoplasty & hernia
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Abdominal Hernia
Keywords: Ventral hernia; Abdominoplasty; Hernioplasty
MeSH Terms: conditions — Hernia, Abdominal; Hernia, Ventral | interventions — Abdominoplasty

STUDY DESIGN:
Intervention Model Description: Repair of ventral hernia with hernioplasty or abdominoplasty.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Concomitant abdominoplasty with ventral hernia repair . (Active Comparator): We do abdominoplasty with concomitant repair of the hernial defect and abdominal wall muscles in the same setting.
  Interventions: Procedure: Abdominoplasty with ventral hernia repair versus ventral hernioplasty.
- Ventral Hernioplasty (Active Comparator): We do hernioplasty with mesh placement for a surgical treatment for ventral hernia.
  Interventions: Procedure: Abdominoplasty with ventral hernia repair versus ventral hernioplasty.

INTERVENTIONS:
Procedure: Abdominoplasty with ventral hernia repair versus ventral hernioplasty. — We do surgical treatment for ventral hernia in the form of hernioplasty with surgical mesh placement or by means of abdominoplasty surgical technique.

SUMMARY:
Comparison between hernioplasty alone versus concomitant abdominoplasty with ventral hernia repair regarding efficacy and post-operative recurrence of hernia.

DETAILED DESCRIPTION:
Ventral hernias are very common and do present a challenge because of the risk of recurrence.

Ventral hernias of the abdomen are defined as a non-inguinal, nonhiatal defect in the fascia of the abdominal wall. Annually, there are about 350,000 ventral hernia operations. The repair of these abdominal wall defects is a common surgery performed by general surgeons. Surgery is typically recommended for individuals with acceptable operative risk, symptomatic hernias, or those at elevated risk of developing complications from a hernia. They can affect an individual's quality of life and can lead to hospitalizations and even death in some cases.[1][2][3] Common causes of acquired ventral hernias include previous surgery causing an incisional hernia, trauma, and repetitive stress on naturally weak points of the abdominal wall. These naturally occurring weak points in the abdominal wall include the umbilicus, semilunar line, ostomy sites, bilateral inguinal regions, and esophageal hiatus. Obesity is a large component of hernias as well because it stretches the fascia of the abdomen causing it to weaken. Specifically, the action of repetitive weight gain and loss leads to weakening.[4] Reported recurrence rates after VHR in the literature vary widely and range from 2.7% to 20% for primary ventral hernia (umbilical and epigastric) to 32-37% for incisional hernia repairs, depending on the series in question. (5) Abdominoplasty can be performed in combination with hernia repair in patients with ventral hernias, especially when associated with large midline ventral hernias, diastasis of recti and the associated laxity and abdominal shape deformity, represent aesthetic and functional problems for the patients. So, the surgical treatment of both pathologies at the same time is highly recommended if the patient's general condition permits. This can be achieved by a comprehensive technique incorporating abdominoplasty performed by a transverse lower abdominal incision into any of the hernia repair techniques.(6) The procedure continues to become increasingly popular, and this is attributed to the increasing rates of obesity and subsequent use of weight loss surgery

Aim(s) of the Research (50 words max):

Is to compare the outcome and efficacy of the combined procedure of (abdominoplasty and hernioplasty) to hernioplasty alone according to rate of post operative recurrence of hernia .

ELIGIBILITY:
Inclusion Criteria:

* Patients with age more than 20 years and less than 60 years old.

Female patients.

Patients having ventral hernias with BM more than 25 kg/m2. Patients with floppy abdomen Patients with divercation of recti Patients with an (ASA) classification of 3 or less with no history of DM or other major comorbidities as cardiopulmonary, hepatic, or renal impairment.Exclusion Criteria:

-

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | Baseline
  Comparison between the two procedures regarding the rate of recurrence within the two patients groups.
Umbilical ischaemic changes | Baseline
  Detection of post operative ishaemia and necrosis of umbilicus as a known complication of abdominoplasty procedure.

IPD SHARING:
Plan to Share IPD: No